CLINICAL TRIAL: NCT04530773
Title: Developing and Validating VR-Enabled Ophthalmic Clinics: A New Paradigm for Visual Function Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, Clinical Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020KYPJ092
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2024-01

CONDITIONS: Visual Health of Virtual Reality

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- GROUP1 (Experimental)
  Interventions: Behavioral: Watch VR movies/ Play VR games
- GROUP2 (Experimental)
  Interventions: Behavioral: Watch VR movies/ Play VR games
- GROUP3 (Experimental)
  Interventions: Behavioral: Watch VR movies/ Play VR games
- GROUP4 (Experimental)
  Interventions: Behavioral: Watch VR movies/ Play VR games
- GROUP5 (Experimental)
  Interventions: Behavioral: Watch VR movies/ Play VR games

INTERVENTIONS:
Behavioral: Watch VR movies/ Play VR games — The healthy individuals will watch VR movies or play VR games with different Physical parameters for 60 minutes.

SUMMARY:
This study aimed to design and validate a VR-based ophthalmic clinic that replicates traditional tests of visual acuity, stereopsis, and contrast sensitivity within an immersive digital environment. Using a rigorously developed system based onprogrammable interfaces, and standardized testing paradigms, we compared VR assessments against gold-standard clinical tools in a cohort of healthy adult participants. Key outcomes included test consistency, correlation, user acceptability, visual fatigue, and time efficiency. Our findings offer evidence for the viability of VR as a platform for remote ophthalmic testing and pave the way for scalable digital eye care delivery.

ELIGIBILITY:
Inclusion Criteria:

* The study included healthy individuals older than 18 years of age with a best-corrected visual acuity (BCVA) of <0.1 logarithm of minimum angle of resolution (logMAR) and no ongoing or prior history of ocular or systemic disease.

Exclusion Criteria:

* The study excluded healthy individuals younger than 18 years of age with a best-corrected visual acuity (BCVA) of >0.1 logarithm of minimum angle of resolution (logMAR) with ongoing or prior history of ocular or systemic disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Accommodative Response | 60 min
  The actual amount of accommodation that exists is measured with a skiascope
AC/A Ratio | 60 min
  The ratio of accommodation convergence to accommodation is measured and calculated by maddox

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Opthalmic Center, Guangzhou, Guangdong, China